CLINICAL TRIAL: NCT03871283
Title: Anticoagulation and Antiplatelet Management During Perioperative Period : a Daily Practice Cohort Prospective Study
Brief Title: Anticoagulation and Antiplatelet Management During Perioperative Period
Acronym: OMAHA
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: OMAHA
Record Dates: First submitted 2019-02-19; First posted 2019-03-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Anticoagulants and Bleeding Disorders
MeSH Terms: conditions — Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
the investigators hypothesize that patients do not understand these therapies, and that they are poorly undertaken. In some cases, the anesthesiologist does not understand correctly the indication of the treatment due to lack of information and therefore does not know how to adapt it to the medical situation.

DETAILED DESCRIPTION:
the investigators hypothesize that patients do not understand these therapies, and that they are poorly undertaken. In some cases, the anesthesiologist does not understand correctly the indication of the treatment due to lack of information and therefore does not know how to adapt it to the medical situation.

the investigators want to investigate these transitions: how were they understood by patients, how were they performed, and how does this affect surgery, postoperative morbidity and mortality?

Anticoagulation for prevention of thromboembolic events will not be studied in this study.

The anesthesia team will not be particularly trained in anticoagulants and antiplatelets management to be close to actual care. In the Hospital the investigators have a guide written in 2013 in order to describe all the cases possible. The "control/ goal group" will be the patients who have undertaken strictly the protocol described for their cases in the guide.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* Able to consent
* Taking anticoagulants or antiplatelet drugs in the long term.

Exclusion Criteria:

* Incapacitated adults
* Minor patients

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patient programed for elective surgery
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Ratio of well treated patient | 30 days
  Ratio of well treated patient

SECONDARY OUTCOMES:
bleeding consequence (volume in mL) | 30 days
  bleeding consequence (volume in mL)
Mortality Consequence | 30 Days
  percentage of death
Blood Test Consequence | 30 Days
  deviation in percentage on INR
Morbidity | 30 days
  percentage of rehospitalisation

CONTACTS AND LOCATIONS:
Overall Officials: Olivier DURANTEAU, Resident, Principal Investigator — ERASME UH
Locations (1):
- ERASME Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Yes
if ask by mail send over
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: at the end of the study during 1 month
Access Criteria: Academic hospital